CLINICAL TRIAL: NCT05968859
Title: Peripheral Limitations in Pulmonary Hypertension and Effects of Muscle Training - The PH Training Trial
Brief Title: A Study of Pulmonary Hypertension Peripheral Limitations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-000705; 1K23HL164901-01A1 (NIH)
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension; Healthy
Keywords: Muscle Training
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Training (Active Comparator): Subjects with PAH will be enrolled to complete baseline study assessments, be randomized to undergo aerobic training for 12 weeks, and then repeat study assessments.
  Interventions: Behavioral: Aerobic Training
- Leg Training (Experimental): Subjects with PAH will be enrolled to complete baseline study assessments, be randomized to undergo leg training for 12 weeks, and then repeat study assessments.
  Interventions: Behavioral: Leg Training
- Healthy Controls (No Intervention): Healthy controls will be enrolled to complete the baseline study assessments for generation of normal reference values for comparison. Healthy controls will not undergo randomized exercise training interventions or repeat assessments.

INTERVENTIONS:
Behavioral: Aerobic Training — Aerobic training will be conducted at 30 minutes 3 times a week using brisk walking with target heart rates goals based on percentage of peak HR reserve (HRR= peak-rest HR) during baseline exercise right heart catheterization (RHC). The target HR will progress over the study period from 50% to 70% of peak HR reserve added to resting HR using the standard Karvonen formula (Goal HR = rest HR + target % of HRR). HR will be monitored using Fitbits to guide training intensity with raw data analyzed using the Fitabase platform to monitor compliance
  Arms: Aerobic Training
Behavioral: Leg Training — Leg training will be performed using assigned ankle weights to perform knee extension while seated. Initial weight assignment will be guided by a protocol driven in-person exercise tolerance test using varying weights to identify the optimal initial and target training weight for each patient based on the 10 repetition maximum weight identified during this test. Leg training weight will begin at 40% of the baseline 10-repetition maximum weight for weeks 1-4 during which time patients will be required to complete 3 sets of 10 repetitions (30 repetitions total) on 3 days per week. For weeks 4-8, 55% of the initial 10-repetition maximum weight will be used for 4 sets of 10 repetitions (40 repetitions total). For weeks 8-12, 70% of the initial 10-repetition maximum weight will be used for 5 sets of 10 repetitions (50 repetitions total).
  Arms: Leg Training

SUMMARY:
The investigators are doing this research study to compare whole body aerobic training with isolated leg training (with weights) and its impact on effectiveness in symptoms and quality of life in patients with Pulmonary Arterial Hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary Arterial Hypertension (PAH) Subjects:

   1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
   2. NYHA Class II-IV
   3. LVEF ≥ 40 % within the preceding year.
   4. No hospitalizations due to heart failure in the preceding 30 days.
   5. No recent initiation of pulmonary vasodilator in the last 60 days
   6. Pulmonary arterial hypertension by right heart catheterization (Mean PA pressure ≥ 20 mmHg with PVR>2 Wood units) with no evidence of heart failure with preserved ejection fraction (exercise PCWP <25 mm Hg).
   7. Symptomatic PAH patients with plan to undergo exercise RHC for reassessment of exertional symptoms
2. Healthy Controls:

   1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
   2. No known diagnosis of heart failure

Exclusion Criteria:

* Myocardial infarction, stroke, hospitalization for heart failure, unstable angina pectoris or transient ischemic attack within 30 days prior to the day of screening.
* Planned coronary, carotid, or peripheral artery revascularization.
* Any other condition judged by the investigator to be the primary cause of dyspnea (such as heart failure due to restrictive cardiomyopathy or infiltrative conditions (e.g., amyloidosis), hypertrophic obstructive cardiomyopathy, anemia, or more than moderate mitral or aortic heart valve disease).
* Wheelchair bound or orthopedic inability to exercise
* Chronic hypoxemia with inability to exercise without oxygen supplementation (PAH Subjects) or need for oxygen supplementation (Healthy Controls)
* Skeletal muscle myopathy
* History of rhabdomyolysis
* Participation in any clinical trial of an approved or non-approved device for the treatment of pulmonary hypertension within 30 days before screening.
* Receipt of any investigational medicinal product within 30 days before screening
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Major surgery scheduled for the duration of the trial, affecting walking ability in the opinion of the investigator.
* Any disorder, including severe psychiatric disorder, suicidal behavior within 90 days before screening, and suspected drug abuse, which in the investigator´s opinion might jeopardize subject´s safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle O2 diffusive conductance (Dm) during supine cycle exercise | Baseline, approximately 12 weeks
  Dm is measured in ml/mm Hg/min during supine cycle exercise

SECONDARY OUTCOMES:
Change in peak O2 consumption (peak VO2) during supine cycle exercise | Baseline, approximately 12 weeks
  Peak VO2 is measured as milliliters of oxygen per kilogram of body weight per minute (ml/kg/min) during supine cycle exercise.
Change in skeletal muscle O2 diffusive conductance (Dm) during single knee-extensor exercise | Baseline, approximately 12 weeks
  Dm is measured in ml/mm Hg/min during single knee-extensor exercise.
Change in maximal mitochondrial respiration | Baseline, approximately 12 weeks
  Measured for the respiratory complexes (complex I+II) per mitochondrial protein content (pmol O2/μg mito/sec) from a quadriceps tissue biopsy.
Change in Quality of Life as measured by the 36-Item Short-Form Survey (SF-36) | Baseline, approximately 8 weeks, approximately 12 weeks
  The SF-36 questionnaire measures quality of life through a range of questions asking about patients physical and mental functioning. The SF-36 has a scale of 0-100 with lower scores indicating more disability and lower quality of life.
Change in Quality of Life as measured by the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) questionnaire | Baseline, approximately 8 weeks, approximately 12 weeks
  PAH-SYMPACT is a PAH-specific patient-reported outcomes instrument that quantifies PAH symptoms and impacts as a measurement of quality of life. The Symptom part is a daily diary that contains 12 items. The respondent is asked to rate each of the items for the past 24 hours. The response options for each item range from 0 " "no [symptom] at all" to 4 "very severe".
Change in Quality of Life as measured by the emPHasis-10 questionnaire | Baseline, approximately 8 weeks, approximately 12 weeks
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items that address breathlessness, fatigue, control, and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Reddy, M.B.B.S, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials